CLINICAL TRIAL: NCT06631573
Title: Prosthetic Complications in Fixed All-On-Four Prosthesis Reinforced with Poly Ether Ether Ketone (PEEK) Versus Cobalt Chromium (Co-Cr) Framework in Completely Edentulous Mandibular Arches. (Randomized Controlled Clinical Trial)
Brief Title: Prosthetic Complications in Fixed All-On-Four Prosthesis Reinforced with Poly Ether Ether Ketone (PEEK) Versus Cobalt Chromium (Co-Cr) Framework
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohannad Alaa Eldin Samy, Assistant lecturer - Prosthodontic department - Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11223
Record Dates: First submitted 2024-09-16; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-12

CONDITIONS: Complete Edentulism
Keywords: all on four , PEEK, Co-Cr, Cobalt Chromium, hybrid prosthesis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed all-on-four prosthesis reinforced with PEEK framework. (Experimental)
  Interventions: Other: fixed all-on-four prosthesis reinforced with PEEK framework.
- Fixed all-on-four prosthesis reinforced with Co-Cr framework (Active Comparator)
  Interventions: Other: Fixed all-on-four prosthesis reinforced with Co-Cr framework

INTERVENTIONS:
Other: fixed all-on-four prosthesis reinforced with PEEK framework. — Prosthetic rehabilitation of mandibular edentulous arches with fixed all-on-four prosthesis reinforced with PEEK framework.
  Arms: Fixed all-on-four prosthesis reinforced with PEEK framework.
Other: Fixed all-on-four prosthesis reinforced with Co-Cr framework — Prosthetic rehabilitation of mandibular edentulous arches with fixed all-on-four prosthesis reinforced with Co-Cr framework
  Arms: Fixed all-on-four prosthesis reinforced with Co-Cr framework

SUMMARY:
Prosthetic complication will be measured for all-on-four fixed prosthesis in the mandibular arch in completely edentulous patients.

DETAILED DESCRIPTION:
Four implants will be placed in the edentulous mandible following all on four surgical protocol. After 3 months as a healing phase, a definitive prosthesis will be fabricated after ensuring the complete osseointegration of all implants. Provisional restorations will be removed, and final impressions will be taken for each patient using addition silicon impression materials. Framework will be constructed using either Cobalt Chromium (Co-Cr) or Poly Ether Ether Ketone (PEEK) according to the randomization process. Jaw relation and try-in will be done to ensure the correct centric relation. Final prosthesis is then screwed to the abutments and the screw hole channels are closed with composite resin restorations. Occlusal adjustments will be done after the delivery and in the subsequent follow up visit. Prosthetic complications (primary outcome) and biological considerations (secondary outcome) will be measured every 3 months along the follow up period which is one year.

ELIGIBILITY:
Inclusion Criteria:

* Any completely edentulous patient (mandible) with an old satisfactory denture requiring an implant-supported restoration.
* Patients aged from 50 to 70, able to sign an informed consent will be considered eligible for this trial.
* Implant sites must allow the placement of four implants.
* Non- heavy Smokers will be included (smoking up to 10 cigarettes/day)
* In case of post-extractive sites, they must have been healed for at least 3-month before being treated in the study.
* Patients with no systemic condition that may interfere with implant placement (e.g., Immunosuppressed or immunocompromised patients, patients under treatment of intravenous amino-bisphosphonates)

Exclusion Criteria:

* Patients with poor oral hygiene and motivation.
* Pregnancy or nursing.
* Drug abusers.
* Psychiatric problems or unrealistic expectations.
* Patients with infection and or inflammation in the area intended for implant placement.
* Patients participating in other studies, if the present protocol cannot be properly adhered to.
* Patients with signs of hyperactive muscles.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Prosthetic complications | one year
  record any prosthetic problem that occurs during the follow up period (such as screw loosening, screw fracture, prosthesis fracture, ....etc.)

SECONDARY OUTCOMES:
Biological considerations | one year
  measure any biological problem in soft tissue around the implants (bleeding on probing, suppuration, .... etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt